CLINICAL TRIAL: NCT06119490
Title: Evaluation of the Efficacy and Safety of Methylprednisolone Combined With the JAK Inhibitors in the Treatment of Toxic Epidermal Necrolysis: Two-arm, Open, Single-center Study
Brief Title: Evaluation of the Efficacy and Safety of Methylprednisolone Combined With the JAK Inhibitors in the Treatment of Toxic Epidermal Necrolysis
Acronym: TEN
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peng Zhang (Other)
Responsible Party: Sponsor-Investigator, Peng Zhang, Investigator, Fujian Provincial Hospital
Organization: Fujian Provincial Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IECFOM-2023-400
Record Dates: First submitted 2023-10-23; First posted 2023-11-07 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Toxic Epidermal Necrolysis
MeSH Terms: conditions — Stevens-Johnson Syndrome | interventions — abrocitinib; Methylprednisolone Hemisuccinate; tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arocitinib-arm (Other): Evaluation of the efficacy and safety of methylprednisolone combined with abrocitinib in toxic epidermal necrolysis. Methylprednisolone 1 mg/kg body weight per day in combination with Arocitinib 200 mg daily.
  Interventions: Drug: Abrocitinib
- Tofacitinib-arm (Other): Evaluation of the efficacy and safety of methylprednisolone combined with tofacitinib in toxic epidermal necrolysis. Methylprednisolone 1 mg/kg body weight per day in combination with tofacitinib 10 mg daily.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Abrocitinib — Solu-Medrol® 1 mg/kg body weight intravenous infusion per day in combination with Arocitinib tablets 200 mg per day for 2 weeks
  Other Names: Solu-Medrol®
  Arms: Arocitinib-arm
Drug: Tofacitinib — Solu-Medrol® 1 mg/kg body weight intravenous infusion per day in combination with Tofacitinib tablets 10 mg per day for 2 weeks
  Other Names: Solu-Medrol®
  Arms: Tofacitinib-arm

SUMMARY:
To evaluate the efficacy and safety of methylprednisolone combined with the JAK inhibitor abxitinib and tofacitinib in the treatment of toxic epidermal necrolysis

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above.
2. Diagnosed with SJS/TEN according to the Registry of Severe Cutaneous Adverse Reactions (RegiSCAR) criteria.
3. Liver and kidney function is within acceptable ranges.
4. Blood parameters, including complete blood count, coagulation function, and platelet count, are within acceptable ranges.
5. Patients must sign an informed consent form, understanding the risks and potential benefits of the treatment.
6. Patients need to be capable of participating in follow-up visits and treatment plans.

Exclusion Criteria:

1. History of allergy to JAK inhibitors.
2. Pregnant or breastfeeding women.
3. Severe infectious conditions.
4. History of central nervous system demyelinating diseases.
5. History of lymphoproliferative diseases.
6. Active and latent tuberculosis.
7. HIV carriers with a CD4+ T cell count lower than (<200/mL).
8. Active HBV/HCV infection.
9. Coagulation disorders or a tendency for thrombosis.
10. Significant abnormalities in blood routine indicators.
11. Liver or kidney dysfunction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Time to Reepithelization | up to 8 week
  duration from initiation of treatment to the point when skin detachment and erosions were no longer observed (negative Nikolsky's sign). Meanwhile, skin islands started to regenerate and replace the damaged superficial epithelia in local skin or mucous lesions (approximately 20% of the maximum BSA).

SECONDARY OUTCOMES:
Adverse events | up to 12 weeks
  The common adverse effects associated with treatments including elevated blood pressure, elevated blood glucose, gastrointestinal bleeding, electrolyte disturbance, and mucocutaneous infections were closely monitored during their hospitalization. All patients in both groups were followed up for 4 weeks to monitor the associated adverse effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, the First Affiliated Hospital of Fujian Medical University., Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided
The results will be published in a peer-reviewed scientific paper and the data sets analyzed in this study can be obtained from the first author.